CLINICAL TRIAL: NCT02672345
Title: Systemic Inflammatory Response Evaluation With the Use of Inhaled Anesthetic Sevoflurane During CPB
Status: Completed | Type: Observational
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Thiago Augusto Azevedo Maranhão Cardoso, MD, Instituto Dante Pazzanese de Cardiologia
Other Study IDs: 4617
Record Dates: First submitted 2016-01-28; First posted 2016-02-03 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Inflammatory Response
Keywords: Sevoflurane; MicroRNAs; Inflammatory Response; Cytokines; Anesthetics, Inhalation; Macrophage Inflammatory Proteins
MeSH Terms: conditions — Respiratory Aspiration | interventions — Sevoflurane

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sevoflurane Group: Group of patients receiving sevorane during extracorporeal circulation period.
  Interventions: Drug: Sevoflurane
- Not Sevoflurane Group: Group of patients who did not receive the sevorane during extracorporeal circulation period.

INTERVENTIONS:
Drug: Sevoflurane — The Sevoflurane Group will receive between 0.7 and 1.5% of sevoflurane CAM only during CPB period. While Not Sevoflurane Group will receive only intravenous anesthetic agents.
  Groups: Sevoflurane Group

SUMMARY:
Cardiac surgery has evolved considerably after the advent of cardiopulmonary bypass (CPB), a feature that allowed more precision and tranquility to the heart surgeon. But their influence on exacerbation of inflammatory response can unbalance the whole homeostasis so happens surgical trauma. The attenuation of the systemic inflammatory response in major surgeries like cardiac surgery for aortic aneurysm appears to represent an important advance in reducing morbidity and mortality of these patients. Some studies suggest that inhaled anesthetics such as sevoflurane appear to play an important role in this control, but the mechanism by which this happens is still unclear. This study has the primary purpose of analyzing from a clinical study sevoflurane inhalation anesthetic can change the inflammatory response induced by CPB, significantly reducing the release of inflammatory markers, especially elastase PMN.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Cardiac Surgery elective of coronary artery bypass graft with cardiopulmonary bypass (CPB)
* The informed consent signature savvy

Exclusion Criteria:

* Use of steroids or anti-inflammatory drugs routine
* Presence of asthma, COPD, autoimmune diseases
* Participation in other clinical studies
* Presence of decompensated heart failures, liver or kidney
* Combined elective surgery (ex .: aneurysm correction + CABG)
* Acute myocardial infarction in the last 30 days
* Unstable angina
* And obesity (BMI> 50kg / m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Will be selected 100 patients who underwent cardiac surgery of coronary artery bypass graft electively in Dante Pazzanese Institute of Cardiology (IDPC).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Reduction of systemic inflammatory response | Through study completion, an average of 1 year
  Cytokines are assayed in both groups at 4 different times in order to check the impact of sevoflurane on the inflammatory response. The first one is the baseline of measurement with which the others are compared and all will be compared within and between groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Thiago Augusto Azevedo Maranhão Cardoso, São Paulo, Brazil

REFERENCES:
- [Derived] Cardoso TAAM, Kunst G, Neto CN, de Ribamar Costa Junior J, Silva CGS, Bastos GM, Borges JB, Hirata MH. Effect of sevoflurane on the inflammatory response during cardiopulmonary bypass in cardiac surgery: the study protocol for a randomized controlled trial. Trials. 2021 Jan 6;22(1):25. doi: 10.1186/s13063-020-04809-x. PMID 33407763